CLINICAL TRIAL: NCT04630652
Title: Immune Modification of Psoriasis by Selective IL-23 Blockade Using Risankizumab
Brief Title: Risankizumab Long-term Remission Study
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jaehwan Kim (Other)
Collaborators: AbbVie (Industry); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor-Investigator, Jaehwan Kim, Instructor in Clinical Investigation, Rockefeller University
Organization: Rockefeller University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JKI-1011; K23AR080043 (NIH)
Record Dates: First submitted 2020-11-09; First posted 2020-11-16 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Psoriasis
Keywords: Psoriasis; Risankizumab
MeSH Terms: conditions — Psoriasis | interventions — risankizumab

STUDY DESIGN:
Intervention Model Description: The interventional study model is to treat moderate-to-severe psoriasis patients with risankizumab for 4 months and analyze pre- and post-treatment skin biopsy samples to (i) identify regulatory immune cell alterations induced by risankizumab administration in the skin of patients whose psoriasis is cleared without recurrence and (ii) develop pre-treatment predictive models for psoriasis patients that anticipate disease clearance and recurrence.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Psoriasis treatment with risankizumab (Experimental): Moderate-to-severe psoriasis treatment with risankizumab for 16 weeks
  Interventions: Drug: Risankizumab-Rzaa; Procedure: Punch biopsies of the skin at baseline visit; Procedure: Punch biopsies of the skin at week 28 visit

INTERVENTIONS:
Drug: Risankizumab-Rzaa — Risankizumab at a dose of 150 mg with injections administered at baseline, week 4 and week 16 following FDA-approved dosage and time periods
  Other Names: SKYRIZI
Procedure: Punch biopsies of the skin at baseline visit — Two 6 mm punch biopsies of the skin at baseline visit
Procedure: Punch biopsies of the skin at week 28 visit — One 6 mm punch biopsy of the skin at week 28 visit

SUMMARY:
Although the newly developed biologics (drugs derived from living cells cultured in a laboratory) are highly effective in controlling psoriasis, all the biologics should be continuously injected to suppress recurrence of the disease. In this regard, the observation in the phase II clinical trial conducted by us (Laboratory for Investigative Dermatology at the Rockefeller University) was groundbreaking that just a single dose of anti-IL-23p19 antibody (risankizumab, trade name: Skyrizi, study drug in this clinical trial) administration produced disease clearance up to 66 weeks in 46% (6 of 13) of patients. However, there is a lack of understanding about immune regulation in human skin induced by anti-IL-23p19 antibody injection, and there is a need to conduct a psoriasis clinical trial for single-cell sequencing immune cells in human psoriasis skin before and after anti-IL-23p19 antibody administration, and to correlate regulatory immune cell alterations with clinical disease progression. The overall objective of the clinical trial is to study regulatory immune cell alterations induced by anti-IL-23p19 antibody administration in psoriasis patients who achieve long-term disease clearance off drugs.

DETAILED DESCRIPTION:
Although the newly developed biologics targeting IL-23/Th17 axis are highly effective in controlling psoriasis, all the biologics should be continuously injected to suppress recurrence of the disease. In this regard, the observation in our phase I psoriasis clinical trial was groundbreaking that just a single dose of anti-IL-23p19 antibody administration produced disease clearance up to 66 weeks in 46% (6 of 13) of patients. Since FoxP3 mRNA levels remained high in posttreatment biopsy specimens of these patients, we hypothesized that IL-23p19 inhibition increased regulatory T-cell levels or function in resolved psoriatic skin. However, there is a lack of understanding about regulatory immune cell promotion by IL-23p19 inhibition in human skin.

Our overall objectives of the study, are to (i) identify regulatory immune cell alterations induced by anti-IL-23p19 antibody administration in the skin of patients whose psoriasis is cleared without recurrence and (ii) develop pre-treatment predictive models for psoriasis patients that anticipate disease clearance and recurrence after short-term anti-IL-23p19 antibody injection. The rationale for this project is that molecular evidence of immune tolerance induction by IL-23p19 inhibition in human skin is likely to offer a strong clinical framework whereby new strategies to prevent recurrence of chronic inflammatory diseases can be developed. In this study, subjects with moderate-to-severe psoriasis will receive FDA-approved anti-IL-23p19 antibody (Generic name: Risankizumab, Product name: SKYRIZI™ or risankizumab-rzaa) up to 4 months following the FDA-approved indications, usage, dosage, and administration in the FDA-approved dosage forms and strengths through week 16, after which, dosing stops.

ELIGIBILITY:
Inclusion Criteria:

* Adult males or females with a diagnosis of plaque psoriasis for at least 6 months.
* Baseline Psoriasis Area Severity Index (PASI) score > 12.
* More than 10% body surface area has plaque psoriasis involvement.
* Willingness to forgo other available psoriasis therapies, live vaccines, and pregnancy during the trial.
* Ability and willingness to provide informed consent and comply with study requirements.

Exclusion Criteria:

* Non-plaque forms of psoriasis.
* Any previous treatment with agents targeting IL-12 or IL-23, including ustekinumab.
* Treatment with biologic agents within previous 3 months prior to visit 0, including adalimumab, etanercept, and infliximab.
* Treatment with immunosuppressive medications, including methotrexate, cyclosporine, oral retinoids, prednisone, or phototherapy within previous 4 weeks prior to visit 0.
* Topical psoriasis treatment within previous 2 weeks prior to visit 0, including topical corticosteroids, vitamin D analogues, retinoids, calcineurin inhibitors, salicylic acid, and coal tar.
* Any investigational study medication within previous 6 months prior to visit 0.
* History of recent or ongoing uncontrolled bacterial, viral, fungal, or other opportunistic infections.
* Positive QuantiFERON-TB Gold test. PPD tuberculin test may be substituted for QuantiFERON-TB Gold test.
* Receipt of a live vaccine (e.g., varicella, measles, mumps, rubella, cold-attenuated intranasal influenza vaccine, and smallpox) in the previous 6 weeks prior to visit 0.
* Females who are pregnant, lactating, planning on pregnancy during the study period, or unwilling to use a medically acceptable method of birth control.
* Severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, pulmonary, cardiac, or neurological disease, or any other medical condition that, in the investigator's opinion, places the participant at risk by participating in this study.
* Any medical history, including laboratory results, deemed by the investigator to be likely to interfere with their participation in the study, or to interfere with the interpretation of the results, or any social condition that, in the opinion of the Investigator, might pose additional risk to the participant or confound the results of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-04-07 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-07-28 (Estimated)

PRIMARY OUTCOMES:
Determination of regulatory immune cell changes induced by risankizumab | week 52
  Changes of regulatory immune cell proportions in total immune cells harvested from the skin biopsy tissues of subjects who have a reduction of 90% or more from baseline in the Psoriasis Area and Severity Index (PASI; range from 0 to 72) at week 12 and also maintain the 90% reduction in PASI at week 52.

SECONDARY OUTCOMES:
Validation of predictive models that anticipate disease recurrence after risankizumab treatment | week 52
  Sensitivity (range from 0 to 100%) and specificity (range from 0 to 100%) of statistical prediction models with single-cell genomic data from the skin biopsy tissues that predict subjects who have a reduction of 90% or more from baseline in the Psoriasis Area and Severity Index (PASI; range from 0 to 72) at week 12 and also maintain the 90% reduction in PASI at week 52.

CONTACTS AND LOCATIONS:
Overall Officials: Jaehwan Kim, MD, PhD, Principal Investigator — The Rockefeller University
Locations (3):
- United States (3):
  - VA Northern California Health Care System, Sacramento, California
  - University of California Davis Medical Center, Sacramento, California
  - The Rockefeller Univesity, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim J, Oh CH, Jeon J, Baek Y, Ahn J, Kim DJ, Lee HS, Correa da Rosa J, Suarez-Farinas M, Lowes MA, Krueger JG. Molecular Phenotyping Small (Asian) versus Large (Western) Plaque Psoriasis Shows Common Activation of IL-17 Pathway Genes but Different Regulatory Gene Sets. J Invest Dermatol. 2016 Jan;136(1):161-172. doi: 10.1038/JID.2015.378. PMID 26763436
- [Background] Kim J, Bissonnette R, Lee J, Correa da Rosa J, Suarez-Farinas M, Lowes MA, Krueger JG. The Spectrum of Mild to Severe Psoriasis Vulgaris Is Defined by a Common Activation of IL-17 Pathway Genes, but with Key Differences in Immune Regulatory Genes. J Invest Dermatol. 2016 Nov;136(11):2173-2182. doi: 10.1016/j.jid.2016.04.032. Epub 2016 May 13. PMID 27185339
- [Background] Kim J, Kim DJ, Ortenzio FS, Dare L, Frank C, Kost RG, Lowes MA. Patients With Psoriasis and Personalized Trade-offs in Treatment Decisions-Lessons Learned From Focus Groups. JAMA Dermatol. 2016 Jun 1;152(6):720-2. doi: 10.1001/jamadermatol.2016.0501. No abstract available. PMID 27028481
- [Background] Kim J, Tomalin L, Lee J, Fitz LJ, Berstein G, Correa-da Rosa J, Garcet S, Lowes MA, Valdez H, Wolk R, Suarez-Farinas M, Krueger JG. Reduction of Inflammatory and Cardiovascular Proteins in the Blood of Patients with Psoriasis: Differential Responses between Tofacitinib and Etanercept after 4 Weeks of Treatment. J Invest Dermatol. 2018 Feb;138(2):273-281. doi: 10.1016/j.jid.2017.08.040. Epub 2017 Sep 18. PMID 28927890
- [Background] Kim J, Krueger JG. Highly Effective New Treatments for Psoriasis Target the IL-23/Type 17 T Cell Autoimmune Axis. Annu Rev Med. 2017 Jan 14;68:255-269. doi: 10.1146/annurev-med-042915-103905. Epub 2016 Sep 23. PMID 27686018
- [Background] Krueger JG, Ferris LK, Menter A, Wagner F, White A, Visvanathan S, Lalovic B, Aslanyan S, Wang EE, Hall D, Solinger A, Padula S, Scholl P. Anti-IL-23A mAb BI 655066 for treatment of moderate-to-severe psoriasis: Safety, efficacy, pharmacokinetics, and biomarker results of a single-rising-dose, randomized, double-blind, placebo-controlled trial. J Allergy Clin Immunol. 2015 Jul;136(1):116-124.e7. doi: 10.1016/j.jaci.2015.01.018. Epub 2015 Mar 11. PMID 25769911
- [Background] Kim J, Lee J, Gonzalez J, Fuentes-Duculan J, Garcet S, Krueger JG. Proportion of CD4+CD49b+LAG-3+ Type 1 Regulatory T Cells in the Blood of Psoriasis Patients Inversely Correlates with Psoriasis Area and Severity Index. J Invest Dermatol. 2018 Dec;138(12):2669-2672. doi: 10.1016/j.jid.2018.05.021. Epub 2018 Jun 8. No abstract available. PMID 29890167
- [Background] Papp KA, Blauvelt A, Bukhalo M, Gooderham M, Krueger JG, Lacour JP, Menter A, Philipp S, Sofen H, Tyring S, Berner BR, Visvanathan S, Pamulapati C, Bennett N, Flack M, Scholl P, Padula SJ. Risankizumab versus Ustekinumab for Moderate-to-Severe Plaque Psoriasis. N Engl J Med. 2017 Apr 20;376(16):1551-1560. doi: 10.1056/NEJMoa1607017. PMID 28423301
- [Background] Lee E, Trepicchio WL, Oestreicher JL, Pittman D, Wang F, Chamian F, Dhodapkar M, Krueger JG. Increased expression of interleukin 23 p19 and p40 in lesional skin of patients with psoriasis vulgaris. J Exp Med. 2004 Jan 5;199(1):125-30. doi: 10.1084/jem.20030451. PMID 14707118
- [Background] Gordon KB, Strober B, Lebwohl M, Augustin M, Blauvelt A, Poulin Y, Papp KA, Sofen H, Puig L, Foley P, Ohtsuki M, Flack M, Geng Z, Gu Y, Valdes JM, Thompson EHZ, Bachelez H. Efficacy and safety of risankizumab in moderate-to-severe plaque psoriasis (UltIMMa-1 and UltIMMa-2): results from two double-blind, randomised, placebo-controlled and ustekinumab-controlled phase 3 trials. Lancet. 2018 Aug 25;392(10148):650-661. doi: 10.1016/S0140-6736(18)31713-6. Epub 2018 Aug 7. PMID 30097359
- [Derived] Kim J, Lee J, Lee J, Kim K, Li X, Zhou W, Cao J, Krueger JG. Psoriasis harbors multiple pathogenic type 17 T-cell subsets: Selective modulation by risankizumab. J Allergy Clin Immunol. 2025 Jun;155(6):1898-1912. doi: 10.1016/j.jaci.2025.02.008. Epub 2025 Feb 18. PMID 39978685